CLINICAL TRIAL: NCT00832208
Title: Open-Label, Sequential Step, Safety and Efficacy Study to Determine the Optimal Single Dose of Ambisome for Patients With Visceral Leishmaniasis
Brief Title: Open-Label, Sequential Step, Safety and Efficacy Study to Determine the Optimal Single Dose of Ambisome for Patients With VL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Addis Ababa University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMBI 0106
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambisome control: (Active Comparator): Ambisome, Total dose 21.0 mg given as 7 x 3mg on days 1,2,3,4,5, and 14 and 21
  Interventions: Drug: Liposomal amphotericin B (Ambisome)
- Ambisome test (Experimental): Single dose Ambisome in sequence(7.5 / 10.0/ 12.5 / 15.0mg)
  Interventions: Drug: Liposomal amphotericin B (Ambisome)

INTERVENTIONS:
Drug: Liposomal amphotericin B (Ambisome) — 21.0 mg/kg total dose. Given iv as 3mg/kg/day on days 1,2,3,4,5, and 14 and 21
  Other Names: Ambisome
  Arms: Ambisome control:
Drug: Liposomal amphotericin B (Ambisome) — liposomal amphotericin b given intravenously as single dose at 7.5 mg/kg increasing to 10, 12.5 and 15.0mg/kg depending on results of interim analyses.
  Other Names: Ambisome
  Arms: Ambisome test

SUMMARY:
This is a phase II/III open, comparative dose trial to find the lowest single dose of AmBisome for the treatment of primary, symptomatic visceral leishmaniasis(VL), in HIV negative patients. In this trial, the minimum effective dose will be determined in a sequential step, dose escalation design, which minimises the number of patients exposed to low, potentially inadequate doses and provides contemporaneous comparative data against the manufacturer's recommended dose schedule in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults and children aged 4 years or older with no upper age limit (in accordance with manufacturer's instructions)
* Acute, symptomatic, VL proven by parasitological examination of splenic aspirate (or bone marrow aspirate) with initial parasite index of at least 2+
* Haemoglobin >4g/dL
* Fever for more than 2 weeks
* Living within reachable distance of the trial site to enable attendance for follow-up visits
* Written informed consent to participate (for children, by parent or guardian)
* HIV negative status

Exclusion Criteria:

* Patients 'in extremis' with signs/symptoms indicative of severe VL
* Patients who have received any anti-leishmanial treatment within the last 6 months
* Patients who have received any investigational (unlicensed) drugs during 6 months before recruitment
* Known underlying chronic disease, such as severe cardiac, pulmonary, renal, or hepatic impairment.
* Renal function tests (serum creatinine) outside the normal range
* Liver function tests more than 3 times the normal range at study entry
* Platelet count less than 40,000/ mm3
* Known alcohol abuse
* Pregnancy or lactation
* Concomitant acute drug usage for malaria and bacterial infection, pneumonia within last 7 days
* Known hypersensitivity to AmBisome or amphotericin B
* Any other condition which may invalidate the trial

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is parasitological clearance with no relapse at 6 months post treatment (ie definitive cure) assessed by clinical status and confirmed by splenic or bone marrow aspiration. | at 6 months post treatment

SECONDARY OUTCOMES:
Parasitological clearance at day 30. | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sisay Yifru, MD, Principal Investigator — Gondar University
Locations (3):
- Ethiopia (2):
  - Gondar, Gonder, Gondar
  - Arba Minch LRTC, Arba Minch
- Kassab Hospital, Kassāb, Gedarif, Sudan

REFERENCES:
- [Derived] Khalil EA, Weldegebreal T, Younis BM, Omollo R, Musa AM, Hailu W, Abuzaid AA, Dorlo TP, Hurissa Z, Yifru S, Haleke W, Smith PG, Ellis S, Balasegaram M, EL-Hassan AM, Schoone GJ, Wasunna M, Kimutai R, Edwards T, Hailu A. Safety and efficacy of single dose versus multiple doses of AmBisome for treatment of visceral leishmaniasis in eastern Africa: a randomised trial. PLoS Negl Trop Dis. 2014 Jan 16;8(1):e2613. doi: 10.1371/journal.pntd.0002613. eCollection 2014. PMID 24454970
- [Derived] Edwards T, Omollo R, Khalil EA, Yifru S, Musa B, Musa A, Wasunna M, Smith PG, Royce C, Ellis S, Balasegaram M, Hailu A. Single-dose liposomal amphotericin B (AmBisome(R)) for the treatment of visceral leishmaniasis in East Africa: study protocol for a randomized controlled trial. Trials. 2011 Mar 6;12:66. doi: 10.1186/1745-6215-12-66. PMID 21375777